CLINICAL TRIAL: NCT04886284
Title: Combination Cefazolin With Ertapenem for Methicillin-susceptible Staphylococcus Aureus Bacteremia (CERT)
Brief Title: Combination Cefazolin With Ertapenem for Methicillin-susceptible Staphylococcus Aureus Bacteremia
Acronym: CERT
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Todd C. Lee MD MPH FIDSA (Other)
Responsible Party: Sponsor-Investigator, Todd C. Lee MD MPH FIDSA, Associate Professor of Medicine, McGill University Health Centre/Research Institute of the McGill University Health Centre
Organization: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2021-7400
Record Dates: First submitted 2021-05-10; First posted 2021-05-14 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Staphylococcus Aureus Bacteremia; Staphylococcus Aureus Septicemia; Staphylococcal Sepsis; Staphylococcus Aureus Endocarditis
Keywords: Staphylococcus aureus; Methicillin-susceptible; Bacteremia
MeSH Terms: conditions — Staphylococcal Infections; Bacteremia | interventions — Ertapenem

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ertapenem (Experimental): Ertapenem 1g IV daily infused over 2 hours x 5 days
  Interventions: Drug: Ertapenem
- Placebo (Placebo Comparator): Saline placebo infused daily over 2 hours x 5 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ertapenem — Adjunctive ertapenem
  Other Names: Invanz
  Arms: Ertapenem
Drug: Placebo — Saline placebo
  Arms: Placebo

SUMMARY:
There is a variety of in vitro, in vivo (animal model), and human case series data which suggests that the addition of ertapenem to cefazolin could improve outcomes in methicillin-susceptible S. aureus bacteremia. No randomized controlled trial has been performed.

This study is an approved sub-study of The Staphylococcus aureus Network Adaptive Platform (SNAP) trial (NCT05137119)

DETAILED DESCRIPTION:
Cefazolin is licensed in Canada for the management of infections due to susceptible Staphylococcus aureus, including bacteremia. It has been commonly used for decades in this disease and, when compared in observational studies to anti-staphylococcal penicillins, has demonstrated reduced mortality.

Nevertheless, in the treatment of methicillin-susceptible S. aureus (MSSA) bacteremia, there remains significant opportunities to improve clinical outcomes. Indeed, S. aureus bacteremia kills more Canadians annually than myeloma, melanoma, renal, ovarian or stomach cancers. Overall mortality approached 18% in a recent Canadian clinical trial performed by our group (Cheng et al, 2020).

The duration of bacteremia, particularly after antibiotherapy is recognized as a major risk factor for mortality. Interventions which reduce the duration of bacteremia, without increasing the frequency of renal failure like gentamicin (Cosgrove et al, 2009) or the combination of vancomycin and flucloxacillin in MRSA (Tong et al, 2020), are among the most promising candidates for larger phase 3 studies designed to impact patient mortality.

Ertapenem is a commonly used antibiotic which has been on the Canadian market for more than 15 years. It is most commonly used in patients with infections caused by extended-spectrum beta-lactamase producing Enterobacteraciae; however, it has a broad spectrum of activity including Gram-positive bacteria such as S. aureus. Indeed, the drug is licensed in Canada for the treatment of complicated skin and soft tissue infections commonly caused by S. aureus.

In S. aureus the carbapenem antibiotics like ertapenem have exceptional affinity to the essential penicillin-binding protein (PBP), PBP1, exceeding even that of the antistaphylococcal β-lactams (Chambers et al, 1990). This complements the relative PBP2 proclivity of cefazolin (Bamberger et al, 2002).

The combination of cefazolin with ertapenem has also been shown to be synergistic in vitro (Sakoulas et al, 2016), in vivo in the mouse and rat models (Sakoulas et al, 2016; Ulloa et al, 2020), and in a small human case series (Ulloa et al, 2020).

Based on this data, there is compelling theory (attack on 2 PBPs), in vitro, in vivo, and human case evidence to support an exploratory phase 2 RCT of cefazolin-ertapenem for the treatment of MSSA bacteremia.

ELIGIBILITY:
The participant must fulfil all inclusion and exclusion criteria for the SNAP Platform (NCT05137119) and also the following inclusion and exclusion criteria to be eligible for this sub-study:

Inclusion Criteria:

1. Adult >=18 years old
2. S. aureus bacteremia within the past 48 hours:

   * with any unknown MRSA status (in centers with <15% prevalence of MRSA in their annual blood cultures) or known negative MRSA screening swab within 90 days OR
   * which has already been shown to be MSSA
3. Current receipt of cefazolin or where it would be clinically appropriate (according to treating ID specialist) to switch to cefazolin as the backbone therapy (open label, non-study drug).

NOTE: Up to an additional 12-24 hours of open label non-study VANCOMYCIN, LINEZOLID or DAPTOMYCIN may be allowed if there is sepsis and clinical concern for MRSA has not been excluded.

Exclusion Criteria:

Clinical:

1. At time of recruitment, the patient has already clinically improved with at least one subsequent negative culture at >24 hours incubation
2. Anaphylaxis to any beta-lactam antibiotic (and any allergy to ertapenem) Polymicrobial bacteremia (not including skin commensals)
3. Known seizure disorder
4. Any receipt of valproic acid
5. Expected mortality within 48 hours
6. Need for critical care resources but "do not resuscitate" status precludes the receipt of critical care
7. Unable to provide informed consent and no available healthcare proxy (with ethics approval for deferred consent in cases of severe illness)

Administrative:

1. Refusal to provide informed consent
2. Refusal of healthcare team to participate
3. No reliable means of outpatient contact (telephone/email/text)
4. Previously enrolled
5. Patients whose isolate is identified as MRSA post-enrollment will be subsequently excluded (see below).

Note that because MSSA is much more common than MRSA in Canada (90% of all S. aureus bacteremia at MUHC, for example, are MSSA and in the presence of a negative MRSA screening swab or unknown MRSA status, this means that the risk of MRSA is less than 5%). We believe time to combination therapy is likely linked to benefit, therefore we will recruit the patients as soon as S. aureus is identified but potentially prior to confirmation the organism is MSSA. Where possible, rapid MRSA detection techniques will be deployed; however with conventional screening this will mean approximately a 12-24 hours delay. Organisms subsequently identified as MRSA will be excluded from the intention to treat analysis and the sample size will be adjusted accordingly to ensure the total enrollment meets study goals.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-05-20 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Clinical success | Day 5
  Composite of: Patient alive, fever resolved, blood cultures negative for S. aureus, systolic blood pressure >=90mmHg not on vasopressors

SECONDARY OUTCOMES:
Blood culture clearance | 30 days
  Time between first positive and first negative blood culture
Clinical improvement | 30 days
  Time to clinical improvement defined as the time until fever resolved, blood cultures sterile, and systolic blood pressure >=90mmHg not on vasopressors in patients who survive to clinical improvement
Length of stay | 90 days
  The time from initial emergency room visit until discharge from hospital in patients discharged alive
All cause-mortality | 90 days
  Death from any cause
C. diff infection | 56 days
  Any C. difficile infection within 56 days
Gram-negative bacteremia | 56 days
  Any Gram-negative bacteremia within 56 days
New colonization with carbapenemase producing organisms | 56 days
  Newly identified colonization with carbapenemase producing organisms to day 56
Valve replacement surgery | 56 days
  Any valve replacement surgery occurring after the initial diagnosis
Recurrent isolation of MSSA from a sterile site | Between Days 6 and 90 inclusive
  Any positive culture of MSSA from a sterile site (blood, cerebral spinal fluid, joint aspirate, bone, etc.) occurring after the end of combination therapy
Seizure | 7 days
  Any clinically identified seizure within 48 hours of discontinuation of combination therapy
Acute Kidney Injury | 7 days
  An increase in serum creatinine to ≥1.5 times baseline OR new requirement for hemodialysis at any time in the first 7 days from randomization

OTHER OUTCOMES:
Health-related quality of life | 90 days
  This will be assessed using the EQ-5D-5L questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Todd C Lee, MD MPH FIDSA, Principal Investigator — Research Institute of the McGill University Health Centre; Emily G McDonald, MD MSc, Principal Investigator — Research Institute of the McGill University Health Centre; Matthew P Cheng, MD, Principal Investigator — Research Institute of the McGill University Health Centre
Locations (5):
- Canada (5):
  - Foothills Medical Centre, Calgary, Alberta
  - Hamilton Health Sciences (Hamilton General Hospital and Juravinski Hospital), Hamilton, Ontario
  - Niagara Health - Niagara Falls Site, Niagara Falls, Ontario
  - Hospital de la Cité de la Sante, Laval, Quebec
  - McGill University Health Centre (Royal Victoria Hospital and Montreal General Hospital), Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ulloa ER, Singh KV, Geriak M, Haddad F, Murray BE, Nizet V, Sakoulas G. Cefazolin and Ertapenem Salvage Therapy Rapidly Clears Persistent Methicillin-Susceptible Staphylococcus aureus Bacteremia. Clin Infect Dis. 2020 Sep 12;71(6):1413-1418. doi: 10.1093/cid/ciz995. PMID 31773134
- [Background] Sakoulas G, Olson J, Yim J, Singh NB, Kumaraswamy M, Quach DT, Rybak MJ, Pogliano J, Nizet V. Cefazolin and Ertapenem, a Synergistic Combination Used To Clear Persistent Staphylococcus aureus Bacteremia. Antimicrob Agents Chemother. 2016 Oct 21;60(11):6609-6618. doi: 10.1128/AAC.01192-16. Print 2016 Nov. PMID 27572414
- [Background] Cosgrove SE, Vigliani GA, Fowler VG Jr, Abrutyn E, Corey GR, Levine DP, Rupp ME, Chambers HF, Karchmer AW, Boucher HW. Initial low-dose gentamicin for Staphylococcus aureus bacteremia and endocarditis is nephrotoxic. Clin Infect Dis. 2009 Mar 15;48(6):713-21. doi: 10.1086/597031. PMID 19207079
- [Background] Bamberger DM, Herndon BL, Fitch J, Florkowski A, Parkhurst V. Effects of neutrophils on cefazolin activity and penicillin-binding proteins in Staphylococcus aureus abscesses. Antimicrob Agents Chemother. 2002 Sep;46(9):2878-84. doi: 10.1128/AAC.46.9.2878-2884.2002. PMID 12183241
- [Background] Chambers HF, Sachdeva M. Binding of beta-lactam antibiotics to penicillin-binding proteins in methicillin-resistant Staphylococcus aureus. J Infect Dis. 1990 Jun;161(6):1170-6. doi: 10.1093/infdis/161.6.1170. PMID 2345297
- [Background] Cheng MP, Lawandi A, Butler-Laporte G, De l'Etoile-Morel S, Paquette K, Lee TC. Adjunctive Daptomycin in the Treatment of Methicillin-susceptible Staphylococcus aureus Bacteremia: A Randomized, Controlled Trial. Clin Infect Dis. 2021 May 4;72(9):e196-e203. doi: 10.1093/cid/ciaa1000. PMID 32667982
- [Background] Tong SYC, Mora J, Bowen AC, Cheng MP, Daneman N, Goodman AL, Heriot GS, Lee TC, Lewis RJ, Lye DC, Mahar RK, Marsh J, McGlothlin A, McQuilten Z, Morpeth SC, Paterson DL, Price DJ, Roberts JA, Robinson JO, van Hal SJ, Walls G, Webb SA, Whiteway L, Yahav D, Davis JS; Staphylococcus aureus Network Adaptive Platform (SNAP) Study Group. The Staphylococcus aureus Network Adaptive Platform Trial Protocol: New Tools for an Old Foe. Clin Infect Dis. 2022 Nov 30;75(11):2027-2034. doi: 10.1093/cid/ciac476. PMID 35717634
- See also: SNAP Platform Registration — https://classic.clinicaltrials.gov/ct2/show/NCT05137119
- See also: SNAP Trial Website — https://www.snaptrial.com.au/